CLINICAL TRIAL: NCT01563861
Title: Determining the Cell of Origin and Prognostic Gene Signatures in SWOG Trials of Diffuse Large B-Cell Lymphoma
Brief Title: S9704-S0014-S0313A Studying Genes in Samples From Patients With Limited or Advanced Diffuse Large B-Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000729157; S9704-S0014-S0313A (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Gene Expression Profiling; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies genes in samples from patients with limited and advanced diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the proportion of the cell of origin subtypes (germinal center B-cell-like [GCB] vs non-GCB) and expression levels of prognostic genes previously identified in diffuse large B-cell lymphoma (DLBCL) in patient biopsy samples from SWOG trials of limited- and advanced-stage DLBCL, and to assess the association between the results and progression-free survival (PFS).
* To assess the association between these marker results and overall survival (OS).

OUTLINE: Archived formalin-fixed paraffin-embedded tissue are analyzed for gene expression profile by quantitative nuclease protection assay (qNPA) and immunohistochemical analyses. Results are then compared with each patient's progression-free survival and overall survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diffuse large B-cell lymphoma - Initial diagnostic tissue block, or 4 unstained slides
* Tissue from patients with limited-stage DLBCL enrolled on SWOG trials treated with cyclophosphamide, doxorubicin hydrochloride, prednisone, and vincristine sulfate (CHOP), and monoclonal anti-CD20 antibody backbone

  * SWOG-S0014
  * SWOG-S0313
* Tissue from patients with advanced-stage DLBCL enrolled on SWOG trials treated with CHOP and monoclonal anti-CD20 antibody backbone

  * SWOG-S9704
  * SWOG-S0433
  * SWOG-S0515
  * SWOG-S0806

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registering to S9704-S0014-S0313 consenting to banking
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 1997-09-15 (Actual); Primary Completion 2008-06-01 (Actual); Study Completion 2013-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of GCB phenotype among limited-stage vs advanced-stage patients | Retrospectively
Differences in PFS between limited- and advanced-stage patients with the GCB and non-GCB phenotypes | Retrospectively
Association between GCB markers and OS | Retrospectively

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O. Persky, MD, Principal Investigator — University of Arizona